CLINICAL TRIAL: NCT01700517
Title: Postoperatory Analgesia After Total Knee Arthroplasty Comparing Femoral and Sciatic-femoral Block
Brief Title: Postoperatory Analgesia After Total Knee Arthroplasty
Acronym: PAINCONTROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Madre Teresa (Other)
Responsible Party: Principal Investigator, Lucio Honorio de Carvalho Junior, PhD, PrincipalInvestigator, PhD, COORDINATOR OF KNEE SURGERY GROUP, ASSOCIATED PROFESSOR, PRINCIPAL INVESTIGATOR, Hospital Madre Teresa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TKR-PAIN CONTROL
Record Dates: First submitted 2012-09-25; First posted 2012-10-04 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: PAIN
Keywords: total knee arthroplasty, analgesia, ultrasonography
MeSH Terms: conditions — Pain; Agnosia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (Sham Comparator): Spinal anesthesia with 0.5% isobaric bupivacaine, in isolation. Punctures in the femoral and popliteal areas were made to mask the femoral and sciatic block, respectively, with no infusion of any medication.
  Interventions: Other: Spinal anesthesia
- Femoral nerve block (Experimental): In addition to the spinal anesthesia, block of the femoral nerve guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. The technique used was femoral area puncture, at the level of the crural fold of skin, with a 0.5% (125mg) ropivacaine associated to 75 mcg of clonidine.
  Interventions: Other: Spinal anesthesia; Other: Femoral nerve block
- sciatic nerves block (Experimental): In addition to the spinal anesthesia and femoral block, the anesthesia of the sciatic nerve at the top of the popliteal fossae was realized, also guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. 0.5% ropivacaine was injected associated to 75mcg clonidine.
  Interventions: Other: Spinal anesthesia; Other: Femoral nerve block; Other: sciatic nerves block

INTERVENTIONS:
Other: Spinal anesthesia — spinal anesthesia
Other: Femoral nerve block — Femoral nerve block
  Arms: Femoral nerve block; sciatic nerves block
Other: sciatic nerves block — sciatic nerves block
  Arms: sciatic nerves block

SUMMARY:
Total knee arthroplasty (TKA) is a worldwide realized procedure, with 600.000 surgeries performed per year in the United States, with a 673% increase estimated until 2030. Functional and pain management improvement is expected in 90% of patients, with 85% of them satisfied after the procedure.

Immediate postoperatory pain control is an important aspect to be considered. Patients submitted to TKA endure pain with variations between 40-80 (according to analog visual scale -AVS - which goes from zero to 100) during the immediate postoperatory, with slow decline in the first 24 hours. Pain classified as severe occurs in 60% and moderated in 30% of patients submitted to TKA during this period of time. Therefore adequate pain management allows an earlier rehabilitation, with a higher satisfaction rate and decrease the hospitalization period.

A multimodal control of pain can be reached by using non-steroidal anti-inflammatory, COX-2 anti-inflammatory inhibitors, peripheral nerve blocks and intra-articular anesthetics injections and decrease use of opioids given of potential collateral effects. Peripheral blockings are associated to the smallest rate of collateral effects and complications when compared to the spinal anesthesia and analgesia controlled by the patients. Studies comparing the effects of the femoral and sciatic-femoral blocking guided by ultrasonography for the analgesia control after TKA were not found.

The objective of this article is to evaluate the effect of femoral and sciatic-femoral block using ultrasonography by the analog visual scale (AVS) of pain in postoperatory of patients submitted to TKA, opioid consumption and complications associated to anesthesics procedures.

DETAILED DESCRIPTION:
Inclusion criteria were considered: Patients with TKA indication, aged from 40 to 90 years, weight between 50 and 100 kg, body mass index between 18 - 36 and patients classified pre-operatory according to the American Anesthesia Association as ASA I or II. Non-cooperative patients, with cognitive incapacity to answer pain VAS, neuromuscular or peripheral neuropathies, chronically using opioid or who didn´t want to take part of the study were taken as exclusion criteria.

The patients were separated in three groups at randomized by a computer program:

Group A - control group - spinal anesthesia, Group B - femoral nerve block + procedure realized in group A and Group C - femoral and sciatic nerves block + procedure realized in group A.

All the anesthetics procedures were realized by the same anesthetist. The standard anesthesia for the procedure was spinal anesthesia with injection of 12 to 15 mg of 0.5% isobaric bupivacaine. Patients of the control group (group A) were submitted to spinal anesthesia with 0.5% isobaric bupivacaine, in isolation. Punctures in the femoral and popliteal areas were made to mask the femoral and sciatic block, respectively, with no infusion of any medication. The patients of the group B received, furthermore the standard anesthesia, the block of the femoral nerve guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. The technique used was femoral area puncture, at the level of the crural fold of skin, with a 0.5% (125mg) ropivacaine associated to 75 mcg of clonidine. For the patients of the group C, in addition to the femoral blocking, the anesthesia of the sciatic nerve at the top of the popliteal fossae was realized, also guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. 0.5% ropivacaine was injected associated to 75mcg clonidine. As an adjuvant for analgesia, all the patients received analgesic and anti-inflammatory permanently in postoperatory, with availability of opioids for rescue if needed. The necessity of its use and eventual complications were registered until hospital discharge.

The pain measurement was realized by the assistant author using a 10 points pain AVS (0, absence of pain, and 10 the worst imaginable pain) both ignoring which group the patient was part of. This measurement was realized during immediate pre-operatory, within 6, 12, 24, 48 hours after surgery.

Details of this study were approved by the Ethical Committee and written informed consent was obtained from each participant prior to the commencement of the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were considered: Patients with TKA indication, aged from 40 to 90 years, weight between 50 and 100 kg, body mass index between 18 - 36 and patients classified pre-operatory according to the American Anesthesia Association as ASA I or II.

Exclusion Criteria:

* Non-cooperative patients, with cognitive incapacity to answer pain VAS, neuromuscular or peripheral neuropathies, chronically using opioid or who didn´t want to take part of the study were taken as exclusion criteria.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LUCIO H CARVALHO, PhD, Principal Investigator — HOSPITAL MADRE TERESA - UNIVERSIDADE FEDERAL DE MINAS GERAIS; EDUARDO F TEMPONI, MD, Study Director — MADRE TERESA´S HOSPITAL
Locations (1):
- Hospital Madre Teresa, Belo Horizonte, Minas Gerais, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 patients submitted to TKA in Madre Teresa´s Hospital between 2011 and 2012 by three authors were enrolled in this prospective, randomized, placebo controlled and double-blinded study after receiving three different types of anesthesia.
Pre-assignment Details: Non-cooperative patients, with cognitive incapacity to understand the AVS, neuromuscular or peripheral neuropathies, chronicle use of opioids or the ones who didn´t want to take part of the study were excluded.
Groups:
- Femoral Nerve Block: In addition to the spinal anesthesia, block of the femoral nerve guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. The technique used was femoral area puncture, at the level of the crural fold of skin, with a 0.5% (125mg) ropivacaine associated to 75 mcg of clonidine.
  Spinal anesthesia : spinal anesthesia
  Femoral nerve block : Femoral nerve block
- Control Group: Spinal anesthesia with 0.5% isobaric bupivacaine, in isolation. Punctures in the femoral and popliteal areas were made to mask the femoral and sciatic block, respectively, with no infusion of any medication.
  Spinal anesthesia : spinal anesthesia
- Sciatic Nerves Block: In addition to the spinal anesthesia and femoral block, the anesthesia of the sciatic nerve at the top of the popliteal fossae was realized, also guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. 0.5% ropivacaine was injected associated to 75mcg clonidine.
  sciatic nerves block : sciatic nerves block
  Spinal anesthesia : spinal anesthesia
  Femoral nerve block : Femoral nerve block
Period: Overall Study
Arm/Group | Femoral Nerve Block | Control Group | Sciatic Nerves Block
Started | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Block | Control Group | Sciatic Nerves Block | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 9 | 21
  >=65 years | 32 | 36 | 31 | 99
Age Continuous [Mean (Standard Deviation); unit: years] | 72 (8.8) | 71.9 (8) | 71.8 (7) | 71.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 34 | 94
  Male | 12 | 8 | 6 | 26
Region of Enrollment [Number; unit: participants]
  Brazil | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Postoperatory Analgesia After Total Knee Arthroplasty Comparing Femoral and Sciatic-femoral Block
Description: The objective of this article is to evaluate the effect of femoral and sciatic-femoral block using ultrasonography by the analog visual scale (AVS) of pain in postoperatory of patients submitted to TKA, opioid consumption and complications associated to anesthesics procedures.
  To assure the double blindness, pain measurement was realized by the assistant author using a 10 points pain analog visual scale (0, absence of pain, and 10 the worst imaginable pain). Patient and researcher did not know at which group patient belongs. This measurement was realized during immediate pre-op, and 6, 12, 24 and 48 hours after surgery. After this the average of pain for each group was analyzed.
Time Frame: 48 HOURS
Population: This sample size was calculated for a fixed effects one-way analysis of variance design. It was assumed that the standard effect size (d) = 0.5, the level of alpha (two-tailed) = 0.05, and power = 0.8, resulting in twenty six patient. The sample was stratified, having 40 patients in each of three groups to compensate for expected dropouts
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Femoral Nerve Block: In addition to the spinal anesthesia, block of the femoral nerve guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. The technique used was femoral area puncture, at the level of the crural fold of skin, with a 0.5% (125mg) ropivacaine associated to 75 mcg of clonidine.
  Spinal anesthesia : spinal anesthesia
  Femoral nerve block : Femoral nerve block
  To assure the double blindness, pain measurement was realized by the assistant author using a 10 points pain analog visual scale (0, absence of pain, and 10 the worst imaginable pain). Patient and researcher did not know at which group patient belongs. This measurement was realized during immediate pre-op, and 6, 12, 24 and 48 hours after surgery. After this the average of pain for each group was analyzed.
- Control Group: Spinal anesthesia with 0.5% isobaric bupivacaine, in isolation. Punctures in the femoral and popliteal areas were made to mask the femoral and sciatic block, respectively, with no infusion of any medication.
  Spinal anesthesia : spinal anesthesia
  To assure the double blindness, pain measurement was realized by the assistant author using a 10 points pain analog visual scale (0, absence of pain, and 10 the worst imaginable pain). Patient and researcher did not know at which group patient belongs. This measurement was realized during immediate pre-op, and 6, 12, 24 and 48 hours after surgery. After this the average of pain for each group was analyzed.
- Sciatic Nerves Block: In addition to the spinal anesthesia and femoral block, the anesthesia of the sciatic nerve at the top of the popliteal fossae was realized, also guided by ultrasonography (Nemio 17 - Toshiba Systems Co. - Japan) and neurosimulation (Stimuplex HNS 12 - Braun - Germany) with 1 Hz stimulus frequency, 1.2 to 0.5 mA energy. 0.5% ropivacaine was injected associated to 75mcg clonidine.
  sciatic nerves block : sciatic nerves block
  Spinal anesthesia : spinal anesthesia
  Femoral nerve block : Femoral nerve block
  To assure the double blindness, pain measurement was realized by the assistant author using a 10 points pain analog visual scale (0, absence of pain, and 10 the worst imaginable pain). Patient and researcher did not know at which group patient belongs. This measurement was realized during immediate pre-op, and 6, 12, 24 and 48 hours after surgery. After this the average of pain for each group was analyzed.
Arm/Group | Femoral Nerve Block | Control Group | Sciatic Nerves Block
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 2 [0 to 10] | 2.8 [0 to 10] | 1.5 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Femoral Nerve Block | Control Group | Sciatic Nerves Block
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
The relative small sample size is one of them. Differences between groups are expected to grow as sample size increases. Despite an improvement in pain control with femoral and sciatic femoral blocks, the morphine consumption was not reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No